CLINICAL TRIAL: NCT02210013
Title: Ethnicity as a Determinant of Ovarian Aging: Differences Between Caucasian and Indian Women
Brief Title: Differences in Ovarian Aging Between Caucasian and Indian Women
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, Juan A Garcia-Velasco, MD, Phd, IVI Madrid
Other Study IDs: MAD-CI-01-2012-01
Record Dates: First submitted 2014-07-29; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Age of the Patients and the Body Mass Index in Both Groups
Keywords: AMH, AFC, aging, ethnicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caucasian women: 200 Caucasian infertile women undergoing their first or second IVF cycle
- Indian women: 200 Indian women undergoing their first or second IVF cycle.

SUMMARY:
The investigators want to carry out a prospective study of 400 infertile Caucasian and Indian women who will undergo a controlled ovarian stimulation for in vitro fertilization (IVF). The investigators will collect data about ovarian reserve markers and also the results after ovarian stimulation in both ethnic groups.The aim is to identify differences in ovarian response after IVF stimulation between both groups.

DETAILED DESCRIPTION:
A total of 200 Caucasian patients and 200 Indian patients who will attend the first or second IVF cycle will be included.

The date we will collect in both groups include the age, the body mass index, and the ovarian reserve markers like the antral follicle count (AFC), the follicle stimulation hormone (FSH) and antimullerian hormone (AMH) serum levels.

The investigators will also determine the number of oocytes retrieved and the metaphase two oocytes in both groups after IVF stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged < 42 years old, with both ovaries present, undergoing a first or second IVF treatment due to male factor, tubal disease or previous failed intrauterine insemination (IUI).

Exclusion Criteria:

* Women diagnosed of polycystic ovary syndrome according to Rotterdam criteria, endometriosis stage III-IV, or previous pelvic inflammatory disease.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Caucasian infertile women and Indican infertile women age < 42 years old, with both ovaries present, undergoing an IVF treatment due to male factor, tubal disease or previous failed IUI.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
AMH levels produced by granulosa cells | day 1
  AMH levels (ng/mL) as well as AFC in both ethnic groups.

SECONDARY OUTCOMES:
Number of oocytes | day 1
  The number of oocytes retrieved as well as the mature oocytes after IVF ovarian stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Iglesias, M.D., Principal Investigator — IVI Madrid; Manish Banker, M.D., Principal Investigator — NOVA IVI; Nalini Mahajan, M.D., Principal Investigator — NOVA IVI; Leyre Herrero, Ph. D., Principal Investigator — IVI Madrid; Antonio Pellicer, M.D., Principal Investigator — IVI VALENCIA; Juan Antonio Garcia-Velasco, M.D., Principal Investigator — IVI Madrid